CLINICAL TRIAL: NCT02080806
Title: Effects of Mechanical Insufflation-exsufflation in Stroke Patients With Dysphagia - Pilot Study
Brief Title: Pilot Study of Efficacy of Mechanical Insufflation Exsufflation in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Sun Im, Assistant Professor, The Catholic University of Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HC 13OISE0066_3; BCMC13AH06 (Other: Bucheon St Marys' Hospital, The Catholic University of Korea)
Record Dates: First submitted 2014-03-05; First posted 2014-03-06 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Stroke; Dysphagia
Keywords: stroke, dysphagia, cough, mechanical insufflation exsufflation
MeSH Terms: conditions — Stroke; Deglutition Disorders; Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mechanical insufflation exsufflation (Active Comparator): Application of cough assist machine as part of the regular physiotherapy
  Interventions: Device: Mechanical Insufflation Exsufflation

INTERVENTIONS:
Device: Mechanical Insufflation Exsufflation — Mechanical Insufflation Exsufflation -Each patient received daily treatments by means of a light-weight, elastic oronasal mask. Treatments were divided between morning and afternoon and were carried out 5 times a week. A total of 20 sessions were carried out by a a trained respiratory therapist.

SUMMARY:
Stroke patients with dysphagia have restrictive lung dysfunction and impaired cough response. This pilot study was performed to determine if Mechanical Insufflation Exsufflation (MIE) therapy can help recover impaired cough function.

DETAILED DESCRIPTION:
Mechanical Insufflation- Exsufflation (MI-E) is an assisted coughing machine that has been proven to be very effective in preventing the deterioration of pulmonary function in patients with degenerative neuromuscular disorders. Impaired airway clearance in stroke patients is associated with increased incidence of aspiration pneumonia.

In this pilot study the investigators attempt to assess the efficacy of MI-E as part of a protocol for patients with dysphagia with impaired cough response.

ELIGIBILITY:
Inclusion criteria Presence of neurogenic dysphagia Presence of impaired cough function

Exclusion criteria Episodes of acute pneumonia or diagnosis of pulmonary embolism at time of enrollment.

Previous history of chronic respiratory dysfunction or other systemic disorders that may impair respiratory function (ex,rheumatoid arthritis, chronic renal disorder, spinal cord injury) Episodes of diaphragm weakness due to peripheral polyneuropathy or phrenic nerve injury Concomitant diagnosis of myopathy, muscular dystrophy, or other neurodegenerative disorders.

Episodes of rib fracture within one year of enrollment. Chronic alcoholism Diagnosis of bullous emphysema Diagnosis of chronic renal failure

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Coughing force as assessed by peak cough flow meter | baseline, 2 weeks

SECONDARY OUTCOMES:
Maximal inspiratory and expiratory pressure | baseline- 2 weeks
Cough force during reflexive cough test | baseline, 2 weeks

OTHER OUTCOMES:
Incidence of pneumonia | baseline 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sun Im, Principal Investigator — The Catholic University of Korea
Locations (1):
- Bucheon St Mary's Hospital, Bucheon-si, South Korea